CLINICAL TRIAL: NCT02661789
Title: Neuropsychobiological Correlates of Sex-steroid Hormone Manipulation in Healthy Women: a Risk Model for Depression
Acronym: GnRHa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gitte Moos Knudsen (Other)
Collaborators: Center for Integrated Molecular Brain Imaging, Copenhagen, Denmak (Other); Rigshospitalet, Denmark (Other); Glostrup University Hospital, Copenhagen (Other); Danish Multiple Sclerosis Center Rigshospitalet (Unknown); Dept. of Clinical Immunology, Rigshospitalet (Unknown)
Responsible Party: Sponsor-Investigator, Gitte Moos Knudsen, Center director of Center for Integrated Molecular Brain Imaging, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GnRHa; H-2-2010-108 (Other: Ethical Committee)
Record Dates: First submitted 2016-01-13; First posted 2016-01-22 (Estimated); Last update posted 2016-01-22 (Estimated); Status verified 2016-01

CONDITIONS: Postpartum Depression; Major Depressive Disorder; Postpartum Psychosis; Menopause; Neurodegeneration; Schizophrenia
Keywords: Mental health; Brain Imaging; Steroid hormones; Serotonin; PET; MRI; fMRI; human; gender; risk model
MeSH Terms: conditions — Depression, Postpartum; Depressive Disorder, Major; Nerve Degeneration; Schizophrenia; Psychological Well-Being; Coitus | interventions — Goserelin; Drug Implants; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GnRHa (Active Comparator): Goserelin 3.6 mg implant
  Interventions: Drug: Goserelin 3.6 mg implant
- Placebo (Placebo Comparator): Injection of saline
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Goserelin 3.6 mg implant — Pharmacologically induced biphasic sex-steroid hormone fluctuation
  Other Names: Zoladex
  Arms: GnRHa
Drug: Placebo — Injection of saline
  Other Names: Saline
  Arms: Placebo

SUMMARY:
The project aimed at identifying neuropsychobiological signatures of pharmacological sex-steroid hormone manipulations in healthy women as a risk model for depression.

The study is a double-blind, randomized, placebo-controlled study. Investigators included 63 healthy female volunteers with regular menstrual cycles between 23 and 35 days. Participants were randomized to active Gonadotrophin-Releasing-Hormone agonist (GnRHa) (goserelin 3.6 mg implant) or placebo (saline injection) intervention, which was initiated in the mid follicular phase (i.e. cycle day 22.6 ±2.5). Sixty women completed follow-up and entered the analyses, except for a few drop outs on some domains. The following domains were addressed at baseline and at follow-up (16±3 days post intervention), (which corresponded to the early ovarian suppression phase of the biphasic hormone response to GnRHa): 1) serotonin transporter binding as imaged by 11CDASB Positron Emission Tomography (PET), 2) functional Magnetic Resonance Imaging (fMRI) emotional processing, 3) fMRI reward processing, 3) rating state fMRI (rsfMRI), 4) structural MRI, 5) Neuropsychology, 6) Psychophysiology, 7) Hypothalamus-Pituitary-Adrenal cortex (HPA)-axis dynamics, 8) Peripheral markers of immunoactive cell responses, 9) Epigenetic factors.

Psychometrics in terms of self reported mental distress and interview based ratings were monitored across the intervention period to monitor potential symptoms of mental distress and psychopathology. Also ovarian hormone responses, peripheral blood markers, and side effects scores were collected across the intervention period.

DETAILED DESCRIPTION:
Aims and hypotheses:

Gender matters in normal brain function as well as in neuropsychiatric disorders. E.g. the vulnerability to mood and anxiety disorders is considerably greater in women. Among other factors, this possibly reflects gender differences in central serotonergic function since dysfunction of serotonergic neurotransmission is critically involved in the pathophysiology of mood and anxiety disorders, schizophrenia, and Alzheimer's disease. In particular, women going through phases in life where sex hormones decline rapidly from high levels or fluctuate, have a higher frequency of severe mood state changes and are more vulnerable to psychiatric disorders, e.g. across the pre to postpartum and menopausal transition. Interestingly, this risk is associated with increased variability of the plasma levels of the sex-hormone estradiol. Therefore, sex-hormone manipulation with a pharmacologically induced biphasic ovarian hormone response serve as a unique opportunity to study how sex-hormone fluctuations provoke mood state changes and increase vulnerability to neuropsychiatric disorders.

In this project investigators aimed at investigating whether sex-hormone manipulation affects: 1. Molecular imaging markers of serotonergic neurotransmission in vivo, 2. Brain structure, architecture and functional connectivity, 3. Stress and inflammatory responses, and 4. Cognitive functions, emotional processing, and information filtering, of importance in the pathophysiology of neuropsychiatric disorders.

Mentally healthy female volunteers were assessed at baseline (i.e cycle day 6.6 ±2.2) and at follow-up (i.e 16.2 ±2.6 days post intervention) in the early ovarian suppression phase af a Gonadotrophin-Releasing-Hormone agonist response in a placebo-controlled, double-blinded design (cohort size aim: N=30x2).

Research in neurobiological correlates of vulnerability related to sex-hormone changes is pivotal to improve the etiological understanding of brain disorders with gender differences in their incidence and/or nature. Such research may contribute to ameliorate fertility treatment, to improve treatment of mood disorders and schizophrenia, and, ideally, shed light on possible preventive strategies in vulnerable phases of women's lives such as the pre- to post-partum and menopausal transition period.

Hypotheses:

Investigators hypothesised that sex-hormone manipulation is associated with the following: 1. Compromised serotonergic neurotransmission, 2. Changes in functional and structural connectivity and lower hippocampal brain volumes and/or markers of decreased neurogenesis, 3. Increased stress reactivity and inflammatory responses, and 4. Changes in neurocognitive functioning and negative bias in emotional processing and information filtering. Investigators further hypothesised that these changes occur in a manner dependent on the magnitude of the estradiol drop from baseline and dependent on symptoms of depressed and anxious mood.

General study design:

The study is a prospective, double-blinded, placebo-controlled, combined within-subject and between-group design of neuropsychobiological changes in response to hormonal down-regulation. The investigation program will be performed at baseline in the mid-follicular phase, at day 5-8 of the menstrual cycle, and in the down-regulated state, 14-19 days after GnRHa intervention.

Participants. Investigators aimed at including 60 healthy female volunteers, in the age range 18-40 years. Group 1 (N=30) will receive sex-hormone manipulation with GnRHa, and group 2 (N=30) will receive placebo (saline injection). The inclusion will be stratified according to a polymorphism in the serotonin transporter promoter region (5-HTLPR).

The investigation program includes functional brain imaging of the serotonin transporter with [11C]DASB PET (6) and fMRI, structural brain imaging, blood measurements of sex-hormone levels, inflammatory and epigenetic biomarkers, characterization of the cortisol awakening response, and psychophysiological measures of information processing, and monitoring of symptoms of mental distress and psychopathology across the intervention period. An initial screening program will secure inclusion of healthy controls only and determine trait parameters such as genotypes, IQ and personality measures.

The study was registered at and approved by the Danish Ethical Committee before participant inclusion under the protocol identification number: H-2-2010-108. All participants gave written informed consent.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women
* Regular menstrual cycles (23 -35 days cycle length)
* No systemic or intrauterine steroid hormone use

Exclusion Criteria:

* Psychiatric disorder (DSM IV Axis I or WHO ICD-10 diagnostic classification).
* Prior or present neurological or other severe medical condition including substance abuse.
* No drug intake suspected to influence results
* Conditions that may increase risk by participating in the study program including ovarian cysts
* Pregnancy during the last year
* Delivery during the last 2 years
* Presently wishing to obtain pregnancy
* Breast feeding
* Not fluent in Danish or severe visual or hearing impairments
* Earlier or present learning disabilities
* Claustrophobia (due to MRI scans)
* Metal implants (excludes MRI)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2011-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in symptoms of depression | Baseline to follow-up 16±3 days after intervention
  Hamilton 17 item score
Changes from baseline in serotonin transporter binding in volumes of interest (VOIs) | Baseline to follow-up 16±3 days after intervention
  PET scan assessed serotonin transporter binding changes
Changes from baseline in fMRI response to emotional faces | Baseline to follow-up 16±3 days after intervention
  fMRI response changes to emotional faces in emotion processing network including amygdala reactivity
Changes from baseline in fMRI response to gambling paradigm | Baseline to follow-up 16±3 days after intervention
  fMRI response changes to reward (monetary win) paradigm in reward processing network
Changes from baseline in rsfMRI changes in functional connectivity | Baseline to follow-up 16±3 days after intervention
  rsfMRI changes in functional connectivity in response to intervention
Changes from baseline in affective cognition (VAMT-24 test) | Baseline to follow-up 16±3 days after intervention
  Neuropsychological (VAMT-24 test) outcomes on affective cognition
Changes from baseline in reaction time | Baseline to follow-up 16±3 days after intervention
  Changes in reaction time
Serial mood fluctuations (SD of total mood disturbance (TMD) score of daily POMS across intervention period) | Intervention start to follow-up 16±3 days after intervention
  Mood fluctuations measured by serial collection of daily POMS
Changes from baseline in hippocampal volume | Baseline to follow-up 16±3 days after intervention
  Hippocampal volumes from structural MRI
Changes in pre-pulse-inhibition (PPI) from baseline | Baseline to follow-up 16±3 days after intervention
  Change in amplitude of the startle response to pulse after pre-pulse warning as measured by EMG in the orbicularis oculi muscle (subtraction of averages across a series of 10 repititions at baseline and at follow-up 16±3 days).
Changes in a set of markers of immunoactivity across study period | Baseline, intervention time, flare-up phase and follow-up
  Cytokines, hsCRP and gene transcript profile markers of
Changes in epigenetic markers of estrogen sensitivity | Baseline to follow-up 16±3 days after intervention
  Epigenetic (methylation) markers
Changes in HPA-axis dynamics (the cortisol awakening response) | Baseline to follow-up 16±3 days after intervention
  The cortical awakening response
Changes in sensorimotor gating (P50 suppression) from baseline | Baseline to follow-up 16±3 days after intervention
  Changes in sensorimotor gating (P50 suppression) from baseline
Changes from baseline in hippocampal microstructure | Baseline to follow-up 16±3 days after intervention
  Hippocampal microstructure from MRI

SECONDARY OUTCOMES:
Changes from baseline in fMRI responses to emotional memory paradigm | Baseline to follow-up 16±3 days after intervention
  Changes in brain activation to fMRI emotional memory paradigm - delayed recall forgetting of word prior to emotional disturbance
Changes from baseline in Cohens perceived stress score | Baseline to follow-up 16±3 days after intervention
  Changes Cohens perceived stress score
Changes in Pittsburg Sleep Quality Inventory (PSQI) | Baseline and 1 time per week until follow-up at 16 ±3 days
  Sleep quality self reported weekly across intervention period
Side effects scores (project specific 15 items questionnaire) | 7, 12 and 30 days post intervention
  Total side effect score across and after intervention period
Changes in SCL-R (Symptom check-list revised) | Baseline and 1 time per week from intervention to follow up at 16±3 days post intervention
  Changes in symptoms of psychopathology across intervention period
Major Depression Inventory (MDI) | Baseline and 1 time per week from intervention to follow up at 16±3 days post intervention
  Changes in self-reported symptoms of depression across intervention period
Changes in profile of mood states (POMS TMD score) | Baseline and 1 time per week from intervention to follow up at 16±3 days post intervention
  Changes in self-reported symptoms of mental distress across intervention period

OTHER OUTCOMES:
Ovarian hormone responses to intervention | Baseline (i.e, cycle day 5-8), intervention time (i.e cycle day 21-23), flare-up phase (i.e, 3-4 days post intervention) and follow-up (i.e.,16±3 days post intervention)
  Ovarian hormone responses to intervention, i.e. concentrations of estradiol, progesterone and testosterone in peripheral blood)

CONTACTS AND LOCATIONS:
Overall Officials: Vibe G Frokjaer, MD, Phd, Principal Investigator — Neurobiology Research Unit
Locations (1):
- Neurobiology Research Unit, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Via database of Center for Integrated Molecular Brain Imaging (Knudsen et al 2016, NeuroImage) data will be available for neuroscience research community contingent on approval by scientific board

REFERENCES:
- [Derived] Mehta D, Rex-Haffner M, Sondergaard HB, Pinborg A, Binder EB, Frokjaer VG. Genome-wide gene expression in a pharmacological hormonal transition model and its relation to depressive symptoms. Acta Psychiatr Scand. 2019 Jul;140(1):77-84. doi: 10.1111/acps.13038. Epub 2019 May 24. PMID 31099405
- [Derived] Fisher PM, Larsen CB, Beliveau V, Henningsson S, Pinborg A, Holst KK, Jensen PS, Svarer C, Siebner HR, Knudsen GM, Frokjaer VG. Pharmacologically Induced Sex Hormone Fluctuation Effects on Resting-State Functional Connectivity in a Risk Model for Depression: A Randomized Trial. Neuropsychopharmacology. 2017 Jan;42(2):446-453. doi: 10.1038/npp.2016.208. Epub 2016 Sep 21. PMID 27649641